CLINICAL TRIAL: NCT04301752
Title: Cognitive Impairment and Neuropsychiatric Manifestations of Neurobrucellosis
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University 13
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Brucellosis
Keywords: Brucellosis, neuropsychiatric manifestations, cognition
MeSH Terms: conditions — Brucellosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurobrucellosis: Brucellosis associated with neuropsychiatric manifestations
  Interventions: Diagnostic Test: MoCA
- Non-neurobrucellosis: Brucellosis not associated with neuropsychiatric manifestations
  Interventions: Diagnostic Test: MoCA

INTERVENTIONS:
Diagnostic Test: MoCA — Cognitive function was assessed by using MoCA score. Cognitive impairment was considered present when MoCA scores were <26. Maximum score is 30.

SUMMARY:
Brucellosis is a common zoonotic infection in many parts of the world including the Mediterranean and Middle Eastern countries.

Neurobrucellosis may develop at any stage of disease and may have widely variable manifestations, including encephalitis, meningoencephalitis, radiculitis, myelitis, peripheral and cranial neuropathies, subarachnoid hemorrhage, and psychiatric manifestations.

DETAILED DESCRIPTION:
Brucellosis is a common zoonotic infection in many parts of the world including the Mediterranean and Middle Eastern countries.

Neurobrucellosis may develop at any stage of disease and may have widely variable manifestations, including encephalitis, meningoencephalitis, radiculitis, myelitis, peripheral and cranial neuropathies, subarachnoid hemorrhage, and psychiatric manifestations.

The aimed is to shed light to the obscure areas of diagnosis in neurobrucellosis and have detailed general and neurologic features

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age with laboratory-confirmed brucellosis

Exclusion Criteria:

* Previous neuropsychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 82 consecutive patients with brucellosis (18 patients with neuropsychiatric manifestations and 64 patients without neuropsychiatric manifestations) were recruited.
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
MoCA s | 24 hours
  Cognitive function was assessed by using MoCA score. Cognitive impairment was considered present when MoCA scores were <26 .

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Young EJ. Brucella species. In: Mandell GL, Bennett JE, Dolin R, eds. Principles and practice of infectious diseases. 7th ed. Philadelphia: Churchill Livingstone, 2010:2921-5.
- [Result] Pappas G, Akritidis N, Bosilkovski M, Tsianos E. Brucellosis. N Engl J Med. 2005 Jun 2;352(22):2325-36. doi: 10.1056/NEJMra050570. No abstract available. PMID 15930423
- [Result] Finn TB. Brucellosis. In: Cohen J, Powderly WG, eds. Infectious diseases. 2nd ed. New York: Elsevier, 2004:1665-9.
- [Result] Eren S, Bayam G, Ergonul O, Celikbas A, Pazvantoglu O, Baykam N, Dokuzoguz B, Dilbaz N. Cognitive and emotional changes in neurobrucellosis. J Infect. 2006 Sep;53(3):184-9. doi: 10.1016/j.jinf.2005.10.029. Epub 2006 May 2. PMID 16647757